CLINICAL TRIAL: NCT06186050
Title: Effects of a High-fat Meal on Exercise-mediated Sympatholysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Philip Millar, Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 23-01-017
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diet, Healthy
Keywords: Functional sympatholysis; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-fat meal with Beetroot Drink (Active Comparator): 2 sausage egg McMuffins and a hashbrown from McDonalds and 10g of beetroot powder mixed in 250 mL cold tap water drink
  Interventions: Dietary Supplement: Beetroot drink
- High-fat meal with Placebo Drink (Placebo Comparator): 2 sausage egg McMuffins and a hashbrown from McDonalds and Mio water flavouring in 250 mL cold tap water. Trace amounts of sugar and sodium were mixed to match the beetroot supplement
  Interventions: Dietary Supplement: Placebo
- Low-fat meal control (Sham Comparator): Kelloggs cornflakes (110g), greek yogurt (400g), skim milk (500 mL), and orange juice (250 mL). Energy-matched to the high-fat meal
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Beetroot drink — Drink containing 10g of beetroot powder in 250 mL cold tap water
  Other Names: Superbeets
  Arms: High-fat meal with Beetroot Drink
Dietary Supplement: Placebo — Mio flavouring in 250 mL cold tap water. Trace amounts of sugar and sodium were added to match the content in the beetroot supplement
  Other Names: Mio
  Arms: High-fat meal with Placebo Drink
Dietary Supplement: Control — Low-fat meal with cornflakes, greek yogurt, skim milk, and orange juice
  Arms: Low-fat meal control

SUMMARY:
The goal of this trial is to examine the effects of a single high-fat meal with or without the co-ingestion of dietary nitrate on exercise-mediated sympatholysis. The main questions it aims to answer are:

1. What are the mechanisms responsible for reduced exercise-mediated sympatholysis following a high-fat meal
2. Can dietary nitrate prevent the declines in exercise-mediated sympatholysis

Participants will be asked to complete three study visits in a randomized order:

1. Low-fat meal
2. High-fat meal
3. High-fat meal plus dietary nitrate

Exercise-mediated sympatholysis will be measured using Doppler ultrasound via a protocol involving rhythmic handgrip exercise and a lower body negative pressure stimulus. Sympatholysis will be assessed before each meal, and at 1, 2, and 3 hours post-prandial.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* Healthy, free of known cardiovascular, metabolic, or musculoskeletal disease

Exclusion Criteria:

* Diagnosed cardiovascular or metabolic disease, injury preventing handgrip exercise, prescription of chronic medications other than oral contraceptives.
* Inability to abstain from drugs (except oral contraceptives), caffeine, alcohol, strenuous physical activity, mouthwash, and multivitamins prior to study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Forearm vascular conductance | Before intervention and 1, 2, 3 hours post-intervention
  Duplex ultrasound of brachial artery
Forearm blood flow | Before intervention and 1, 2, 3 hours post-intervention
  Duplex ultrasound of brachial artery
Systolic and Diastolic Blood Pressure | Before intervention and 1, 2, 3 hours post-intervention
  finger plethysmography

SECONDARY OUTCOMES:
Plasma levels of Norepinephrine | Blood collected before intervention and 1, 2, 3 hours post-intervention. Blood frozen at -80 degrees Celsius and analyzed at later date
  ELISA kit
Plasma levels of Nitrate/Nitrite concentration | Blood collected before intervention and 1, 2, 3 hours post-intervention. Blood frozen at -80 degrees Celsius and analyzed at later date
  ELISA kit
Blood Glucose concentrations | Blood collected before intervention and 1, 2, 3 hours post-intervention. Blood analyzed immediately after collection at each time point
  Blood glucose monitor
Plasma levels of Triglycerides | Blood collected before intervention and 1, 2, 3 hours post-intervention. Blood frozen at -80 degrees Celsius and analyzed at later date
  Triglyceride assay kit

CONTACTS AND LOCATIONS:
Overall Officials: Philip Millar, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph - Human Cardiovascular Physiology Laboratory, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No